CLINICAL TRIAL: NCT05168332
Title: The Influence of Patellar Taping Combined with Isometric Strength Training on Pain, Muscle Strength, and Functional Performance in Individuals with Patellofemoral Pain Syndrome.
Brief Title: The Effect of Patellar Taping and Isometric Strength Training on Quadriceps Strength with Patellofemoral Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S.Hasan
Record Dates: First submitted 2021-12-12; First posted 2021-12-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Patello Femoral Syndrome
Keywords: Patello-femoral pain syndrome; pain; strength; Maximum voluntary Isometric contraction (MVIC).
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Experimental group Control group
Who Masked: Participant
Masking Description: single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental(Group A): patellar taping combined with isometric strength training (Experimental): The experimental group (Group A): patellar taping with isometric strength training for six weeks.
  Interventions: Behavioral: patellar taping combined with isometric strength training; Behavioral: sham patellar taping combined with isometric strength training
- Control group (Group B): sham patellar taping combined with isometric strength training. (Sham Comparator): Control group (Group B): sham patellar taping combined with isometric strength training for six weeks.
  Interventions: Behavioral: patellar taping combined with isometric strength training; Behavioral: sham patellar taping combined with isometric strength training

INTERVENTIONS:
Behavioral: patellar taping combined with isometric strength training — patellar taping combined with isometric strength training
Behavioral: sham patellar taping combined with isometric strength training — sham patellar taping combined with isometric strength training

SUMMARY:
Patellofemoral pain syndrome is one of the most common young adult female complaints, caused by changes in the patellofemoral joint's physical and biomechanical properties. This study compared the Short-term effects of patellar taping combined with isometric contraction of quadriceps muscle strengthening at 900 or 600 knee angles on quadriceps strength and functional performance in a female patient with patello-femoral pain syndrome (PFPS)

DETAILED DESCRIPTION:
Quadriceps muscle strength Pain intensity Knee function

ELIGIBILITY:
Inclusion Criteria:

* knee pain for at least eight weeks that was aggravated by activities such as descending and ascending stairs, squatting, and running.
* knee pain with a positive J sign (lateral tilt of patella)
* more symptomatic and mal align knee included in case of bilateral involvement and a sign of patellar malalignment on the radiograph.

Exclusion Criteria:

* History of knee fracture
* Patella dislocation
* knee deformity (e.g., genu varum)
* Knee Flexion contracture
* Ligament/meniscal injuries,
* NSAID or intra-articular injection, or knee Osteo arthritis.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength | 6 weeks
  Knee extensors (Maximal Voluntary Isometric Contraction) strength (STN) test at 60, and 90 degrees angles
Pain intensity | 6 weeks
  investigated for their current intensity of pain on a Visual analogue scale 0 to 10 scale.
Knee function | 6 weeks
  Knee function will be assessed using the validated Kujala Anterior Knee Pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan, PhD, Principal Investigator — Associate Professor, Majmaah University
Locations (1):
- Rehabilitation center, Majmaah University, Al Majma'ah, Al Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasan S. The effect of patellar taping combined with isometric strength training on pain, muscle strength, and functional performance in patients with patellofemoral pain syndrome: a randomized comparative study. PeerJ. 2025 May 12;13:e19381. doi: 10.7717/peerj.19381. eCollection 2025. PMID 40376557